CLINICAL TRIAL: NCT00703196
Title: HPV Clearance by Folic Acid Supplementation (FACT for HPV)
Brief Title: Folic Acid Clinical Trial for the Prevention of Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000579360; UAB-F060511015; UAB-IRB0000196
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2014-01

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; human papilloma virus infection; low-grade squamous intraepithelial lesion; high-grade squamous intraepithelial lesion; atypical squamous cells of undetermined significance; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Papillomavirus Infections; Squamous Intraepithelial Lesions; Atypical Squamous Cells of the Cervix; Uterine Cervical Dysplasia | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral folic acid pill once daily for 12 months in the absence of unacceptable toxicity or any other adverse effects.
  Interventions: Dietary Supplement: folic acid
- Arm II (Placebo Comparator): Patients receive oral placebo once daily for 12 months in the absence of unacceptable toxicity or any other adverse effects.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: folic acid — Given orally once daily
  Arms: Arm I
Other: placebo — Given orally once daily
  Arms: Arm II

SUMMARY:
RATIONALE: Supplements, such as folic acid, may stop or delay the development of cervical cancer in women infected with human papillomavirus.

PURPOSE: This phase II trial is studying how well folic acid supplements work in preventing cancer in women infected with human papillomavirus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effects of folic acid supplementation on clearance of human papilloma virus (HPV) 16 and other specific types of HR-HPV and on prevention of the progression of ≤ cervical intraepithelial neoplasia (CIN) 1 lesions (not true preneoplastic lesions) to CIN ≥ 2 (true neoplastic lesions) by conducting a 12-month double-blind randomized placebo-controlled trial with 5 mg of folic acid/day.

Secondary

* Evaluate whether the clearance of HPV 16 and other specific HR-HPV types and the progression of cervical lesions (≤ CIN 1 to CIN ≥ 2) is modified by lower levels of circulating and/or cervical cell folate, presence of micronuclei or global DNA hypomethylation in cervical cells, presence of integrated vs episomal HPV 16, or a high HPV 16 viral load in cervical cells at the enrollment.

OUTLINE: This is a single center study. Patients are stratified according to multivitamin use (yes vs no) and smoking status (smoker vs nonsmoker). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral folic acid pill once daily for 12 months in the absence of unacceptable toxicity or any other adverse effects.
* Arm II: Patients receive oral placebo once daily for 12 months in the absence of unacceptable toxicity or any other adverse effects.

All patients complete a diet, physical activity, and a risk factor questionnaire at the enrollment visit (0-month) and at 4, 8, and 12 month visits (a total of 4 visits). Fasting blood samples for assessing circulating concentrations of micronutrients (folate, vitamins B12, A, E, C, and total carotenes) and exfoliated cervical cell samples for assessing HPV are collected at all 4 visits. Anthropometric measures are taken at all study visits. A colposcopically directed biopsy is taken at the 0-month visit and at the 12-month visit to assess the histological diagnoses of cervical lesions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Received care at the Health Departments in Alabama and with an abnormal pap result, including any of the following:

  * Atypical squamous cells of undetermined significance (ASCUS)
  * ASCUS, cannot exclude high-grade lesion (ASCUS-H)
  * Low-grade squamous intraepithelial lesion
  * High-grade squamous intraepithelial lesion
* Referred to University of Alabama at Birmingham (UAB) Highlands Clinic for further colposcopic examination by Ob/Gyn physicians
* Tested positive for human papilloma virus (HPV) 16 and diagnosed with ≤ cervical intraepithelial neoplasia (CIN) 1 lesions at the 0-month visit

  * With or without concurrent infections with other HR (High Risk) HPV types (HPV 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, and 68)
* Not diagnosed with true preneoplastic lesions of the cervix based on a colposcopically directed biopsy

PATIENT CHARACTERISTICS:

* Not pregnant
* Willing to take study pills, keep scheduled follow-up study visits, or communicate with study personnel about changes in contact information during the study period
* No prior diagnosis or treatment for colon polyps or breast lumps

PRIOR CONCURRENT THERAPY:

* No prior treatment for cervical cancer or precancerous condition
* No prior surgeries involving the cervix
* No concurrent antifolate medications such as methotrexate, sulfasalazine or phenytoin
* No concurrent or planned consumption of 400 μg or more of a folic acid supplement on a regular basis
* Not involved in any other clinical trial

Ages: 19 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2007-03; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clearance of HPV 16 and other coexisting HR-HPV and incidence of CIN ≥ 2 | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Chandrika J. Piyathilake, PhD, MPH, Study Chair — University of Alabama at Birmingham
Locations (1):
- UAB Comprehensive Cancer Center, Birmingham, Alabama, United States